CLINICAL TRIAL: NCT03699215
Title: Ensayo clínico, Fase III, Aleatorizado, Prospectivo, unicéntrico, Doble Ciego y Controlado Con Placebo, Para Estimar la Eficacia y Seguridad Del Levosimendan Intravenoso, en Las Primeras 24 Horas Tras la Angioplastia Primaria, en Pacientes Con síndrome Coronario Agudo Con elevación Del Segmento ST
Brief Title: Clinical Trial in Patients Who Have Suffered a Heart Attack and Who Have Undergone Catheterization Treated With Levosimendan
Acronym: LEVOCEST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LEVOCEST
Record Dates: First submitted 2018-09-27; First posted 2018-10-09 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2020-08

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): solution for intravenous infusion, with similar organoleptic characteristics than active treatment.
  Interventions: Drug: Placebos
- levosimendan (Experimental): Concentrate for solution for perfusion. Pack with a 5 ml vial
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan — Upon arrival of the patient in the Coronary Unit, he will receive, in a randomized and double-blind manner, the 24-hour infusion of Levosimendan, without a loading dose, at a dose of 0.1 μg / kg / min or placebo. If the initial dose is tolerated and a greater hemodynamic effect is needed, the infusion rate can be increased to 0.2 micrograms / kg / min. The dose of Levosimendan infusion can be reduced to 0.05 μg / kg / min in case of clinical intolerance or systolic hypotension <90 mmHg.
  Arms: levosimendan
Drug: Placebos — continuous perfusion of 0.1 micrograms / kg / min for 24h. If the initial dose is tolerated and a greater hemodynamic effect is needed, the infusion rate can be increased to 0.2 micrograms / kg / min.
  Arms: placebo

SUMMARY:
The disease under study is acute coronary syndrome with ST segment elevation, defined as patients presenting chest pain of anginal characteristics of more than 20 minutes of duration, with changes in the electrocardiogram consisting of ST segment elevation of 1 mm in two contiguous limb leads or 2 mm in two contiguous leads precordial. In a review carried out on patients treated in the investigator center with SCACEST, invetsigators found that, in a cohort of 250 patients, 85% of them presented alterations Segments of left ventricular contractility at 4 months after the acute episode. To verify that the Levosimendan administration reduces that percentage, at least 65%, investigators require to include in the study 83 patients in the experimental group and 83 in the control group, for a power of 80% and a confidence level of 95%. Assuming 10% of lost patients, it is required to include in the study 92 patients in the experimental group and 92 patients in the group control .

DETAILED DESCRIPTION:
The patients will be included randomly, until the calculated sample size is completed. A recruitment period of 12 months is estimated from the beginning of the study. From the date of inclusion of the first patient, the final duration of the study will be 1.5 years.

The study will end when performing the last cardio-resonance and echocardiography that should be performed 6 months after the inclusion of the last patient in the study.

Upon arrival of the patient at the Coronary Unit, he will receive, in a randomized and double-blind manner, without a loading dose, the 24-hour infusion of Levosimendan, or placebo.

The continuous infusion of levosimendan 0.1 micrograms / kg / min will be administered during 24h. If the initial dose is tolerated and a greater hemodynamic effect is needed, the infusion rate can be increased to 0.2 micrograms / kg / min. The dose of Levosimendan infusion can be reduced to 0.05 μg / kg / min in case of clinical intolerance or systolic hypotension <90 mmHg.

Continuous perfusion of the placebo 0.1 micrograms / kg / min will be administered for 24h. If the initial dose is tolerated and a greater hemodynamic effect is needed, the infusion rate can be increased to 0.2 micrograms / kg / min. The dose of infusion of the placebo can be reduced to 0.05 μg / kg / min in case of clinical intolerance or systolic hypotension <90 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes who come to CHUC.
* Age between 18 and 85 years old.
* Symptoms of STEMI over 30 minutes and less than 12 hours of evolution.
* ST segment elevation of >= 1 mm in two contiguous limb leads or >= 2 mm in two contiguous precordial leads.
* Patients agreed to participate in the study and have signed the informed consent.
* The same patient may not be included more than once.

Exclusion Criteria:

* Killip IV class in a situation of cardiogenic shock or with TAM values below 65 mmHg of pressure.
* Patients that have suffered a previous heart attack.
* Patients who are being administered amines.
* Patients that do not have segmental disorders of contractility in left ventriculography.
* Mental circumstance that makes you unable to participate in the study.
* Patients that refuse to participate in the study and that they do not sign the informed consent.
* Severe renal impairment (creatinine clearance <30ml / min)
* Severe hepatic insufficiency - (prothrombin activity rate <40%).
* History of Torsades de Pointes.
* Acute respiratory distress
* Allergy to levosimendan or some of its components
* Anemia (hemoglobin <8g / dl)
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2018-11-17 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Size of acute myocardial infarction | 30 days after acute episode
  percentage myocardium infarct/ left ventricle ventricle

SECONDARY OUTCOMES:
measurement of Biochemical parameters function | first 24 hours
  troponine, creatinkinase, creatinkinase-MB
electrocardiogram parameters | 1 hour after primary angioplasty
  Residual ST segment deviation
MAJOR CARDIAC EVENTS | 6 months after angioplasty
  need of revascularitation or cardiac death

CONTACTS AND LOCATIONS:
Locations (1):
- UICEC, San Cristóbal de La Laguna, S/C de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No